CLINICAL TRIAL: NCT05860764
Title: Vascular Amputee Physical Performance Qualitative (VAmPP-Q) Study: Exploratory Study Investigating Perceptions and Experience of Physical Performance and Physical Assessment of Vascular Amputees Using Performance Based Outcome Measures
Brief Title: Vascular Amputee Physical Performance Qualitative (VAmPP-Q) Study
Acronym: VAmPP-Q
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0873
Record Dates: First submitted 2022-11-01; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-11

CONDITIONS: Vascular Disease, Peripheral; Amputation; Physical Disability
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vascular amputees and healthcare professionals: participants who have undergone an amputation due to peripheral arterial disease and healthcare professionals who treat these participants

SUMMARY:
Background:

Peripheral arterial disease (PAD) is the main cause of amputation to the lower limb within the UK, affecting over 20% of adults older than 70 years.

After an amputation, individuals often use a wheelchair and do not walk with a prosthetic limb. This is due to them experiencing: older age, muscle weakness, pain, other health conditions limiting ability to exercise eg. heart problems.

Healthcare professionals assess physical function with Physical Performance Based Outcome Measures (PerBOMs). A PerBOM requires an individual to complete tasks that are part of their day to day life e.g. walking or balance.

PerBOMs are used with for:

* Setting goals with patients
* Assessing how patients respond to treatment/rehabilitation
* Predicting if patients are likely to use a prosthetic limb in the future

Previous research shows most of the available PerBOMs are suitable an amputee who walks with a prosthetic limb. However, most vascular amputee patients cannot benefit from these assessments.

Therefore, based on this evidence we have developed a new PerBOM to help manage vascular amputees who do not walk with a prosthetic limb.

Methods:

Qualitative interviews and focus groups with amputee individuals and healthcare professionals who treat them. Approaching individuals who have or will undergo an amputation to their leg due to PAD. Approaching healthcare professionals through professional networks.

Interviews and focus groups will take place face to face or remotely by telephone/video conferencing, lasting approximately 1-2 hrs.

In the interview or focus group, the researcher will explain and show individuals a video of the new PerBOM and explore their opinions qualitatively on this new PerBOM.

All audio will be recorded, written up and analysed. All findings will be presented at scientific conferences.

This study has been developed with patients and public involvement.

ELIGIBILITY:
Vascular amputee group:

Inclusion criteria

* Undergone major lower limb amputation due to peripheral arterial disease and/or diabetes at any time point
* or
* Planned date for major lower limb amputation within 1 week of consent due to peripheral arterial disease and/or diabetes

Exclusion criteria

* Has/will undergo a minor amputation only
* Amputation due to alternative aetiology
* No plan for amputation to lower limb
* Unable to communicate or write in English
* Lacking capacity to consent to research study
* >1 weeks or unspecified date for amputation surgery
* <18 years

Healthcare professional group:

Inclusion criteria

• Healthcare professional currently working with vascular amputees. Healthcare professional defined as qualified professional background e.g. HCPC, NMC or GMC registered or non-qualified professional background e.g. healthcare support worker

Exclusion criteria

* No experience of working with vascular amputee patients
* Unable to speak or write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 groups of participants in one cohort
  * participants who have undergone an amputation due to peripheral arterial disease, 'vascular amputees'
  * healthcare professionals that work with vascular amputees in clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
qualitative theme identification | baseline
  qualitative themes will be identified after data collection through qualitative interviews and focus groups and thematic analysis has taken place

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Sciences, University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No